CLINICAL TRIAL: NCT06747715
Title: Minimally Invasive Post-Traumatic Craniofacial Soft Tissue Regeneration: Validation of Safety and Efficacy of Staged Approach Using Autologous Fresh Fat Grafting Followed by Autologous Cryopreserved Fat Grafting
Brief Title: Autologous Fresh Fat Grafting Followed by Autologous Cryopreserved Fat Grafting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Endowed Chair of Plastic Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24080145
Record Dates: First submitted 2024-11-21; First posted 2024-12-24 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Facial Defect

STUDY DESIGN:
Intervention Model Description: The therapeutic intervention is a two stage surgical procedure (with a third stage biopsy for research purposes in this trial) in which a primary traumatic or post-surgical craniofacial deformity is treated first with autologous fat grafting using freshly harvested adipose tissue. A second fat grafting procedure is performed at 3.0 months after the first procedure using autologous adipose tissue that had been cryopreserved during the first procedure.
  Facial volume and appearance will be scored by 4 blinded observers (2 physicians and 2 lay-observers) from standardized photographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Intervention (Experimental): The therapeutic intervention is a two stage surgical procedure (with a third stage biopsy for research purposes in this trial) in which a primary traumatic or post-surgical craniofacial deformity is treated first with autologous fat grafting using freshly harvested adipose tissue. A second fat grafting procedure is performed at 3.0 months after the first procedure using autologous adipose tissue that had been cryopreserved during the first procedure.
  Interventions: Procedure: Serial Fat Grafting Fresh followed by Cryopreserved Fat

INTERVENTIONS:
Procedure: Serial Fat Grafting Fresh followed by Cryopreserved Fat — The therapeutic intervention is a two stage surgical procedure (with a third stage biopsy for research purposes in this trial) in which a primary traumatic or post-surgical craniofacial deformity is treated first with autologous fat grafting using freshly harvested adipose tissue. A second fat grafting procedure is performed at 3.0 months after the first procedure using autologous adipose tissue that had been cryopreserved during the first procedure.

SUMMARY:
The goal of this clinical trial is to validate the safety and effectiveness of a two-stage approach for minimally invasive craniofacial soft tissue reconstruction using autologous fat grafting in wounded service members and veterans. The main questions it aims to answer are:

1. Will treating subjects with post-traumatic craniofacial deformities using fresh fat grafts, followed by a second treatment 3 months later with cryopreserved fat stored at -80°C, improve facial tissue regeneration and appearance?
2. How do volume retention and tissue health change between fresh and cryopreserved grafts in humans?
3. How do factors such as cellular composition of the graft, patient demographics, and medical conditions (including diabetes, tobacco use, medications, age, and BMI) affect fat graft volume retention and overall outcomes?

Researchers will compare results from the second-stage cryopreserved fat grafting to fresh fat grafting to assess outcomes like volume retention, patient recovery, and cost reduction.

Participants will:

Undergo an initial fat grafting procedure. Have additional fat harvested and cryo-stored for use in a second-stage procedure.

Receive the cryopreserved fat in a later stage without the need for a second fat harvest.

Receive small test injections behind each ear for later analysis. Provide data on demographics and medical conditions for correlation with outcomes.

DETAILED DESCRIPTION:
Craniofacial injuries are common among wounded service members, with 22.7% to 39% of battle injuries affecting the cranio-maxillofacial region. Restoring appearance requires precise soft tissue reconstruction. This proposal aims to address that need using a minimally invasive approach that uses the patient's own tissue, building on previous successful DoD-funded clinical trials.

Autologous fat grafting (AFG) is a common, minimally invasive procedure used in plastic surgery to restore facial volume. In a prior department of defense funded trial, the study investigators demonstrated its safety and effectiveness for repairing traumatic craniofacial deformities. However, about 37% of the grafted fat is reabsorbed during early healing, requiring multiple procedures for optimal results. The donor site harvest is the main source of discomfort, time, and cost in these procedures.

The study investigators propose improving this process by harvesting extra fat during the first procedure, cryo-storing it, and using the preserved fat for a second stage without needing another harvest. This approach will be validated using outcome measures from prior work. Additionally, the investigators are working with a commercial partner to advance a low-cost kit for cryo-storing fat at medical facilities, including military treatment centers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent,
* Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 3 and 150 cc of lipoaspirate (the patient's own fat, collected through liposuction). This may include patients who have not had craniofacial surgical procedures, as well as those who have undergone surgical procedures and have remaining deformities (post-surgical deformities).
* Be at least 3 months post-injury or most recent surgery, so that acute edema (swelling) is resolved.
* Volume defects (facial injury) are covered by intact skin and do not communicate with oral cavity or sinuses.
* The three-dimensional geometry of the volume defects (facial injury) would allow for treatment with fat grafting.
* Has sufficient donor tissue, as assessed on physical exam, to graft deformity and cryostore an equal amount of adipose (fat) tissue.
* Willing and able to comply with follow up examinations, including radiographic studies (i.e. CT scans)

Exclusion Criteria:

* Age less than 18 years.
* Inability to provide informed consent.
* Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: A second facial injury, that will not be treated by the study, that includes this type of defect, will not necessarily exclude the patient from participating).
* Active infection anywhere in the body.
* Systemic disease or medical condition that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
* History of radiation to the areas intended for treatment or the graft harvest site
* Medications that would significantly impact wound healing, such as immunosuppressive agents, chronic steroid treatment, or chemotherapy, or medications/allergies that would pose a risk to anesthesia or the planned procedures.
* Active narcotic abuse (presents a variable for pain logs).
* Known coagulopathy (increased risk of bleeding/delay in forming blood clots).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Facial volume and appearance scale | The key timepoint is 3 months post-graft. The difference between the Facial Volume and Appearance Scale scores from the Pre-treatment baseline to the 3-months post-1st treatment, for each subject, will be generated.
  This is a validated visual 3-point grading scale that will be scored by 4 blinded observers (2 physicians and 2 lay-observers) from standardized photographs The definitions for each of three points on the scale are listed here: a score of 1 means: for baseline grading of a given facial aesthetic region assessed there is an obvious contour defect that would benefit from volume fill. For post-treatment grading, no discernable improvement from baseline. A score of 2 means: for a given facial aesthetic region with a history of a traumatic deformity and treatment of the deformity according to the study protocol, there is a discernable improvement in the contour defect from baseline which does not yet approximate the contralateral side (if uninjured) or represent a normal appearance. A score of 3 means: for a given facial aesthetic region there is a normal appearance and/or close to matching contralateral structure (if uninjured).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From intervention to the final study visit (3 months post 2nd treatment, or approximately 6 months after initial intervention)
  Incidence of adverse events will be counted, as well as a subscore for those adverse events that are considered related to the study intervention.
Change in facial injury volume from Pre to Post CT Scans- within each subject- High resolution Computed Tomography with 3D reconstruction (CT) will be performed. | Facial volume analysis of the injured area will be calculated from the individual CTs, comparing from each subject's pretreatment baseline to the final study visit (3 months post 2nd treatment, or approximately 6 months after initial intervention)
  Craniofacial fine cut CT with 3D reconstruction & volume analysis. 5 CTs of the face will be done on each subject. The first scan will be pre-procedural and will serve as a baseline. All CT scans will be done on a 64-slice scanner (LightSpeed, GE Healthcare), using collimation of 0.625mm and slice interval of 0.3mm, resulting in approximately 50% overlap between adjacent slices. kVp, mA, and FOV will be optimized to the subject, but will approximately be kVp=120; mA=320, FOV=18cm. Soft tissue and bone kernels will be employed. These images will be volumetrically reformatted into coronal and sagittal planes for confirmation of findings. Additionally, surface-rendered volumetric reformats will be created emphasizing both bony structures and soft tissues. Images will be reviewed by a dedicated head and neck radiologist with 25 years of experience in CT of the face.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, Principal Investigator — University of Pittsburgh; Patsy Simon, BS, RN, CCRC, CCRA, ACRP-PM, Study Director — Director, Operations and Administration
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No